CLINICAL TRIAL: NCT03773848
Title: Hook Plate vs Tightrope in Fixation of Fracture Distal Third Clavicle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, David Mounir Kamal Ibrahim, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hook plate vs Tightrope
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Fracture Clavicle

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A- hook plate (Experimental): All participants will have an Open Reduction Internal Fixation (ORIF). The affected upper limb will be temporarily fixed by a sling after admission. The patients will be placed in a beach-chair position in an orthopaedic theatre. The operated side will be prepped and draped and a transverse incision will be made over the fracture site. The fracture ends will be identified, reduced and fixed with hook plate. X-ray was applied to check the grade of reduction before the operation is completed.
  Interventions: Procedure: Open Reduction Internal Fixation (ORIF)
- B- tightrope (Experimental): All participants will have an Open Reduction Internal Fixation (ORIF). The affected upper limb will be temporarily fixed by a sling after admission. The patients will be placed in a beach-chair position in an orthopaedic theatre. The operated side will be prepped and draped and a transverse incision will be made over the fracture site. The fracture ends will be identified, reduced and fixed with tightrope. X-ray was applied to check the grade of reduction before the operation is completed.
  Interventions: Procedure: Open Reduction Internal Fixation (ORIF)

INTERVENTIONS:
Procedure: Open Reduction Internal Fixation (ORIF) — Open Reduction Internal Fixation (ORIF) of fracture lateral third clavicle by hook plate & tightrope

SUMMARY:
to compare the clinical & radiological outcomes of hook plate & tightrope fixation in fracture of lateral third clavicle.

DETAILED DESCRIPTION:
Adult clavicle fractures account for 4% to 10% of fractures. Distal clavicle fractures occurs in 25% to 30% of all clavicle fracture.The management of fractures of the distal clavicle has been a matter of debate in literature. Neer in 1968 suggested a new classification and proposed general treatment guidelines . Type I and type III fractures are generally treated non-operatively. For type II fractures, surgical management is the treatment of choice .There are numerous operative techniques reported in the past. The methods of surgical treatment could be summarised as follows:

1. Fixation in terms of K-wires and different pins such as the Steinmann pin, and Knowles pin. This fixation could also be augmented with concomitant tension band wires
2. Coracoclavicular indirect fixation with the use of screws, suture anchors, Dacron graft or Mersilene tape
3. Open reduction and clavicular plate fixation with the use of different plate systems such as the Balser plate,locked plate,hook plate, etc.

Different surgical techniques have their own advantages and disadvantages With more than 20 techniques described so far, no single fixation is ideal and perfect. There is still no consensus regarding the best surgical method to fix these fracture ,the investigators choose two of the most common of these methods and evaluate & compare best radiological & clinical outcomes of both.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 16 years old) including both sexes.
* Acute fractures within 3 weeks of injury.
* Isolated & closed fractures.

Exclusion Criteria:

* Pathological fracture of distal clavicle.
* Deteriorated general health.
* Previous history of dysfunction with the affected shoulder.
* Incomplete medical records or lost to follow up.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of limb function this change will be assessed using Disabilities of the Arm, Shoulder and Hand (DASH) Score as limb function will be expected of some movement limitation at 6 weeks and no limitations to be at 6 months | at 6 weeks & 6 months post-operatively.
  The DASH is a self-administered questionnaire that consists of thirty core questions and an optional additional eight questions assessing work and sports and/or performing arts activities. Each individual item is scored on a 5-point Likert scale, with lower scores correlating to minimal impairment and higher scores indicating more impairment. The cumulative DASH score is scaled from 0 to 100, with higher scores indicating more disability

SECONDARY OUTCOMES:
Fracture Healing | at 6 weeks & 6 months post-operatively.
  Radiological evaluation of the fracture by using antero-posterior and axillary views x-ray
Blood loss | Intra-operatively
  Recording of the blood loss amount during surgery in milliliters.
Radiation time | Intra-operatively
  Calculation of the exposure time to radiations during surgery in minutes.
Skin condition | at 6 weeks
  Evaluation of skin condition of the surgical incision by clinical inspection

REFERENCES:
- [Background] Flinkkila T, Heikkila A, Sirnio K, Pakarinen H. TightRope versus clavicular hook plate fixation for unstable distal clavicular fractures. Eur J Orthop Surg Traumatol. 2015 Apr;25(3):465-9. doi: 10.1007/s00590-014-1526-9. Epub 2014 Sep 9. PMID 25200315
- [Background] Haque S, Khan A, Sharma A, Sundararajan S. Technical tip: tightrope fixation of neer type II distal clavicle fracture supported by a case series. Pol Orthop Traumatol. 2014 Mar 27;79:19-22. PMID 24675020
- [Background] Lee W, Choi CH, Choi YR, Lim KH, Chun YM. Clavicle hook plate fixation for distal-third clavicle fracture (Neer type II): comparison of clinical and radiologic outcomes between Neer types IIA and IIB. J Shoulder Elbow Surg. 2017 Jul;26(7):1210-1215. doi: 10.1016/j.jse.2016.11.046. Epub 2017 Jan 26. PMID 28131682
- [Background] Yan HW, Li L, Wang RC, Yang Y, Xie Y, Tang J, Shi ZY. Clinical efficacies of coracoclavicular ligament reconstruction using suture anchor versus hook plate in the treatment of distal clavicle fracture. Orthop Traumatol Surg Res. 2017 Dec;103(8):1287-1293. doi: 10.1016/j.otsr.2017.07.006. Epub 2017 Aug 8. PMID 28801112